CLINICAL TRIAL: NCT03723967
Title: Multicenter Prospective Single Arm Phase II Study Evaluating Efficacy & Safety of Durvalumab With Carboplatin/Paclitaxel as First Line Treatment in Patients With Recurrent/Metastatic SCCHN Not Eligible to Standard Chemotherapy
Brief Title: FRAIL-IMMUNE (GORTEC 2018-03) - Combination of Durvalumab With Carboplatin/Paclitaxel
Acronym: FRAIL-IMMUNE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ET18-023 FRAIL-IMMUNE
Record Dates: First submitted 2018-10-18; First posted 2018-10-30 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2022-09

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
Keywords: Squamous Cell Carcinoma of the Head and Neck; Recurrent / metastatic SCCHN; Frail patients; GORTEC
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Recurrence | interventions — durvalumab; Carboplatin; Paclitaxel

STUDY DESIGN:
Intervention Model Description: Multicenter, prospective, single arm phase II study (a run-in tolerance study will be first performed on a limited number of patients: maximum 9)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Durvalumab with Carboplatin/Paclitaxel (Experimental): Combination of Durvalumab with Carboplatin/Paclitaxel as first line treatment in patients with recurrent/metastatic SCCHN not eligible to standard chemotherapy
  Interventions: Drug: Durvalumab with Carboplatin/Paclitaxel

INTERVENTIONS:
Drug: Durvalumab with Carboplatin/Paclitaxel — Durvalumab associated with Carboplatin / Paclitaxel as first line treatment in patients with recurrent/metastatic SCCHN not eligible to standard chemotherapy
  Other Names: Combination of Durvalumab with Carboplatin/Paclitaxel

SUMMARY:
The primary objective of the phase II trial is to determine the efficacy and safety of a combination of Durvalumab with the Carboplatin/Paclitaxel as first line treatment in patients with recurrent/metastatic SCCHN not eligible to standard chemotherapy.

DETAILED DESCRIPTION:
For recurrent or metastatic Squamous Cell Carcinoma of the Head and Neck (SCCHN), the standard first-line treatment is chemotherapy by cisplatin-fluorouracil and cetuximab which allows a median overall survival of 10.1 months. Due to its toxicity, this combination could be proposed only to patients younger than 70 years, good PS (ECOG PS0 or PS1) and adequate renal function.

In routine practice it is estimated that the proportion of eligible patients is about two third. One third of patients were ineligible to first-line chemotherapy by cisplatin-fluorouracil-cetuximab. Among them, 25% due to PS2 and the others for various reasons (older than 70 years, renal insufficiency….). For these ineligible patients, an alternative chemotherapy should be proposed. The carboplatin-paclitaxel scheme with weekly paclitaxel is safe for poor population and demonstrated efficacy in head and neck cancers with overall survival varying from 4.9 months to 12.8 months in first line. The response rate varies from 20% to 52% and is about 25% in our experience. Even for frail patients it should be a safe and active treatment.

Nivolumab, a monoclonal antibody targeting PD1 demonstrated survival benefit compared with chemotherapy in patients with SCCHN who progressed after platinum-based first line (median OS of 7.5 months versus 5.1 months and 12-month OS rate of 36.0% versus 16.6%). Safety data confirm these antibodies are of interest in a population of frail patients. Only 58.9% of patients experienced treatment-related adverse events with nivolumab arm and 13% of grade 3/4. Durvalumab, an anti-PDL1 antibody is currently tested in SCCHN with promising results.

Head and neck cancers are rapidly progressive and due to the delayed action of immunotherapy, and the recent demonstration that immunotherapy with anti-PD1 or anti-PDL1 can be responsible of hyperprogression, patients will probably benefit from addition of chemotherapy to immunotherapy, mostly for patients unfit for cisplatin-fluorouracil because their poor condition is often related to the cancer and a rapid response is needed.

This trial proposes to study the addition of Durvalumab to chemotherapy in first line treatment for frail patients with recurrent/metastatic SCCHN.

Prior to this evaluation, a run-in tolerance study in a limited number of patients to ensure that the experimental treatment combination is safe.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years at the time of study entry;
2. Histological or cytological confirmation of the diagnosis of Squamous Cell Carcinoma of the Head and Neck;
3. Primary tumor located in one of the following : oral cavity, larynx, oropharynx or hypopharynx (NB: sinuses and nasopharynx locations are not allowed; isolated cervical lymphnodes with unknown primary site may be discussed with the coordinating investigator on a case by case basis)
4. Archival tumor sample available at the time of inclusion with sufficient material to achieve the translational research program. Archival material must have been collected 3 months before inclusion at the latest, unless a new tumor sample must be collected.
5. Disease must be in metastatic (Stage IVc) or recurrent setting;
6. Documented progression of measurable disease as per the RECIST 1.1 (NB: in case of a single metastatic lesion, the tumor size must be > 20mm to allow tumor biopsy)
7. Patients must be ineligible to standard therapies, including cisplatin. Ineligibility is defined as at least one of the following criteria:

   * Creatinine clearance (CrCl) : 40 < CrCl < 60ml/min
   * Any severe comorbidity rendering the patient ineligible to standard chemotherapy, as per investigator's judgment.
8. Eastern Cooperative Oncology Group performance status of 0, 1 or 2
9. Must have a life expectancy of at least 12 weeks
10. Body weight > 30Kg;
11. Adequate organ and marrow function as defined below:

    * Hemoglobin ≥ 9.0 g/dl
    * Absolute Neutrophils Count (ANC) ≥ 1.5 x 109/L
    * Platelet count ≥ 100 x 109/L
    * Creatinine clearance ≥ 40 ml/min using the following appropriate formulae:

      * Cockroft-Gault formula for female : 0.85 x weight (Kg) x (140-age) / 72 x serum creatinine (mg/dL)
      * Cockroft-Gault formula for male : weight (Kg) x (140-age) / 72 x serum creatinine (mg/dL)
      * MDRD for patients older than 65 years: 186.3 x (serum creatinine (µmol/L / 88.4) -1.154 x Age -0.203 x (0.742 if female) x (1.212 if black patient [African origin]).
    * AST/ALT ≤2.5 x institutional upper limit of normal unless liver metastases are present, in which case it must be ≤5 x ULN
    * Serum total bilirubin ≤ 1.5 x ULN (in the absence of Gilbert's syndrome)
    * Coagulation panel : INR or PT ≤ 1.5 x ULN
12. Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

    * Women <50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
    * Women ≥50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).
13. Patient (male or female) using a highly effective contraception as defined in appendix 9 during the study treatment period and until 6 months after the last administration of carboplatin and/or paclitaxel or until 90 days after the last administration of durvalumab, whichever is longer. Prior to dispensing study drugs, the investigator must confirm and document the patient's (and his/her partner) use of highly effective contraceptive methods, dates of negative pregnancy tests, and confirm the patient's understanding of the teratogenic potential of study drugs.
14. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
15. Covered by a medical insurance.
16. Signed and dated informed consent document indicating that the patient has been informed of all the pertinent aspects of the trial prior to enrolment

Exclusion Criteria:

1. History of another primary malignancy except for:

   * Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of IP and of low potential risk for recurrence
   * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
   * Adequately treated carcinoma in situ without evidence of disease
2. Prior anticancer therapy in metastatic or recurrent setting In case patient received neoadjuvant or adjuvant anti-cancer treatment, it must have been completed for at least 6 months prior to study drugs initiation and patient must have no unresolved toxicity NCI CTCAE Grade ≥2 with the exception of alopecia, vitiligo and laboratory values defined as inclusion criteria.

   Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the coordinating investigator.

   Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab may be included only after consultation with the coordinating investigator.
3. Any previous treatment with a PD1 or PD-L1 inhibitor, including durvalumab.
4. Patient whom tumor lesion is hemorrhagic or at risk of bleeding
5. Patient whom disease progressed within 6 months after the start date of the previous chemotherapy (faster progressors)
6. Symptomatic or active leptomeningial or parenchymal brain metastases. Patients whose brain metastases have been treated may participate provided they show radiographic stability (defined as 2 brain images, both of which are obtained after treatment ot the brain metastases; these Imaging scans should both be obtained at least 4 weeks apart and show no evidence of intracranial progression). In addition, any neurologic symptoms that developed either as a result of the brain metastases or their treatment must have resolved or be stable either, without the use of steroids, or are stable on a steroid dose of <=10mg/day of prednisone or its equivalent and anticonvulsant for at least 14 days prior to the start of treatment.
7. Active or prior/history of disease/medical condition listed below:

   * Inflammatory or interstitial lung disease
   * Documented autoimmune or inflammatory disease (including inflammatory bowel disease [e.g., Crohn's disease, ulcerative colitis], systemic lupus erythematosus, sarcoidosis syndrome or Wegener syndrome, granulomatosis with polyangitis, Grave's disease, rheumatoid arthritis, hypophysitis, uveitis, etc) within the past 2 years except for autoimmune hypothyroidism on a stable dose of thyroid supplementation and patients with type 1 diabetes mellitus on a stable dose of insulin.

   Note: Subjects with alopecia, vitiligo, psoriasis not requiring systemic treatment (within the past 2 years) or chronic skin condition that does not require systemic therapy, are not excluded, as well as patients without active disease in the last 5 years (after consultation with the study physician) and patients with celiac disease controlled by diet alone.
   * Mean QT interval corrected for heart rate (QTc) ≥470 ms using Fredericia's Correction.
   * Clinically significant cardiac disease or congestive heart failure > New York Heart Association (NYHA) class 2. Patients must not have unstable angina (anginal symptoms at rest) or new-onset angina within the last 3 months or myocardial infarction within the past 6 months.
   * History of primary immunodeficiency
   * Allogeneic organ transplantation
   * Documented hypersensitivity to the active substance or excipient of the study drugs
   * Any uncontrolled intercurrent illness including, but not limited to:

     * Ongoing or active infection, including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and tuberculosis testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
     * Active peptic ulcer disease or gastritis,
     * Active bleeding diatheses including any subject known to have evidence of acute risk,
     * Serious chronic gastrointestinal conditions associated with diarrhea
   * Any psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the subject to give written informed consent
8. Current or prior use, or need for the following concomitant medications/interventions not permitted during the study treatment period :

   * Any concurrent chemotherapy or radiotherapy treatment to more than 30% of the bone marrow or with a wide field of radiation within 4 weeks of the first dose of study drug (except palliative radiotherapy on a non-target lesion after discussion with the coordinating investigator), immunotherapy, biologic or hormonal therapy for cancer treatment, other than any stated in the protocol (Note: concurrent use of hormonal therapy for non-cancer-related conditions (e.g. hormone replacement therapy) is acceptable)).
   * Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab including, but not limited to systemic corticosteroids at doses exceeding 10 mg/day of prednisone or equivalent, methotrexate, azathioprine, and TNF-α blockers. Use of immunosuppressive medications for the management of investigational product-related AEs or in subjects with contrast allergies is acceptable.
   * Phenytoin given in a prophylactic intent
   * Receipt of live attenuated vaccine within 30 days prior to the first dose of IP (Note: Patients, if enrolled, should not receive live vaccine whilst receiving IP and up to 30 days after the last dose of IP).

     * Strong inhibitors and inducers of CYP3A4
     * Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of IP. Note: Local surgery of isolated lesions for palliative intent is acceptable.
9. Participation in another clinical study with an investigational product during the last 28 days prior to first study drug administration
10. Pregnant or breastfeeding women (Women of childbearing potential are required to have a negative serum pregnancy test within 72 hours prior to study treatment start. A positive urine test must be confirmed by a serum pregnancy test).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2019-05-16 (Actual); Primary Completion 2020-05-16 (Actual); Study Completion 2024-03-09 (Actual)

PRIMARY OUTCOMES:
Evaluation of efficacy and safety of Durvalumab with the Carboplatin/Paclitaxel as first line treatment in patients with recurrent/metastatic SCCHN not eligible to standard chemotherapy | 12 months after study treatment initiation
  Number of patients still alive 12 months after the first study drug administration (overall survival)

SECONDARY OUTCOMES:
Progression-Free Survival | 12 months after study treatment initiation
  Defined as the time from the date of the first study drug administration to the date of first documented progression or death due to any cause
Time to Treatment Failure | 12 months after study treatment initiation
  Defined as the time from the date of inclusion to the date of permanent study treatment discontinuation
Overall survival | Up to 36 months
  Defined as the time from the date of inclusion to the date of death due to any cause
Objective Response Rate | 12 months after study treatment initiation
  Defined as the proportion of patients with a best overall response of Complete or Partial Response
Best Response Rate | 12 months after study treatment initiation
  Defined as proportion of patients who achieve a best response of CR, PR, SD or PD
Duration of response | 12 months after study treatment initiation
  Defined as the time from the date of first documented response (CR or PR) to the date of the first documented subsequent progression or death due to any cause
Quality of life using European Organisation for Research and Treatment of Cancer (EORTC) questionnaire | 12 months after study treatment initiation
  Using the EORTC QLQ-C30 (Quality of Life Questionnaire) - Scale range: 1 (better outcome) to 4 (worse outcome) for 28 variables and from 1 (better outcome) to 7 (worse outcome) for 2 variables
Quality of life using European Organisation for Research and Treatment of Cancer (EORTC) questionnaire | 12 months after study treatment initiation
  Using the EORTC QLQ-H&N35 questionnaire (Quality of Life Questionnaire) - Scale range: 1 (better outcome) to 4 (worse outcome) for 30 variables and from 1 (better outcome) to 2 (worse outcome) for 5 variables
Tolerance profile: Incidence of treatment emergent adverse events and serious adverse events | 12 months after study treatment initiation
  Incidence of Treatment Emergent Adverse Events, Serious Adverse Events (SAE) and death assessed according to the NCI-CTC AE version 5

OTHER OUTCOMES:
Determination as predictive & prognostic factors of efficacy: Time to recurrence | Inclusion, Day 1 cycle 2 (each cycle is 28 days), First documented radiological progression
  Time to recurrence in patients with localized disease at diagnosis.
Determination as predictive & prognostic factors of efficacy : Site of recurrence | Inclusion, Day 1 cycle 2 (each cycle is 28 days), First documented radiological progression
  Site of recurrence (in or outside a previous irradiation field for patients who have previously received radiation therapy)
Determination as predictive & prognostic factors of efficacy: Level of expression of PD-L1 | Inclusion, Day 1 cycle 2 (eachy cycle is 28 days), First documented radiological progression
  Determined by immunohistochemistry (archival formalin fixed paraffin embedded tumor sample)
Determination as predictive & prognostic factors of efficacy: Level of expression of p16 | Inclusion, Day 1 cycle 2 (each cycle is 28 days), First documented radiological progression
  Determined by immunohistochemistry (archival formalin fixed paraffin embedded tumor sample)embedded tumor sample)
Determination as predictive & prognostic factors of efficacy: Level of HPV for patients presenting an oropharynx tumour and a tumor with a positive p16 | Inclusion, Day 1 cycle 2 (each cycle is 28 days), First documented radiological progression
  Determined by immunohistochemistry (archival formalin fixed paraffin embedded tumor sample)
Optional outcome: Immune infiltrate assessment: CD3 analysis | Inclusion, Day 1 cycle 2 (each cycle is 28 days), First documented radiological progression
  Determined by multiIF (archival formalin fixed paraffin embedded tumor sample)
Optional outcome: Immune infiltrate assessment: CD8 (T cells) analysis | Inclusion, Day 1 cycle 2 (each cycle is 28 days), First documented radiological progression
  Determined by multiIF (archival formalin fixed paraffin embedded tumor sample)
Optional outcome: Immune infiltrate assessment: CD20 analysis | Inclusion, Day 1 cycle 2 (each cycle is 28 days), First documented radiological progression
  Determined by multiIF (archival formalin fixed paraffin embedded tumor sample)
Optional outcome: Immune infiltrate assessment: CD38 analysis | Inclusion, Day 1 cycle 2 (each cycle is 28 days), First documented radiological progression
  Determined by multiIF (archival formalin fixed paraffin embedded tumor sample)
Optional outcome: Immune infiltrate assessment: IgG analysis | Inclusion, Day 1 cycle 2 (each cycle is 28 days), First documented radiological progression
  Determined by multiIF (archival formalin fixed paraffin embedded tumor sample)
Optional outcome: Immune infiltrate assessment: NKp46 analysis | Inclusion, Day 1 cycle 2 (each cycle is 28 days), First documented radiological progression
  Determined by multiIF (archival formalin fixed paraffin embedded tumor sample)
Optional outcome: Immune infiltrate assessment: FOXP3 | Inclusion, Day 1 cycle 2 (each cycle is 28 days), First documented radiological progression
  Determined by multiIF (archival formalin fixed paraffin embedded tumor sample)
Optional outcome: Immune infiltrate assessment: CD4 analysis | Inclusion, Day 1 cycle 2 (each cycle is 28 days), First documented radiological progression
  Determined by multiIF (archival formalin fixed paraffin embedded tumor sample)
Optional outcome: Immune infiltrate assessment: CD8 analysis | Inclusion, Day 1 cycle 2 (each cycle is 28 days), First documented radiological progression
  Determined by multiIF (archival formalin fixed paraffin embedded tumor sample)
Optional outcome: Immune infiltrate assessment: Treg analysis | Inclusion, Day 1 cycle 2 (each cycle is 28 days), First documented radiological progression
  Determined by multiIF (archival formalin fixed paraffin embedded tumor sample)
Optional outcome: Immune infiltrate assessment: NK analysis | Inclusion, Day 1 cycle 2 (each cycle is 28 days), First documented radiological progression
  Determined by multiIF (archival formalin fixed paraffin embedded tumor sample)
Optional outcome: Immune infiltrate assessment: Monocytes analysis | Inclusion, Day 1 cycle 2 (each cycle is 28 days), First documented radiological progression
  Determined by multiIF (archival formalin fixed paraffin embedded tumor sample)
Optional outcome: Immune infiltrate assessment: DC analysis | Inclusion, Day 1 cycle 2 (each cycle is 28 days), First documented radiological progression
  Determined by multiIF (archival formalin fixed paraffin embedded tumor sample)
Optional outcome: Mutation of genes | Inclusion, Day 1 cycle 2 (each cycle is 28 days), First documented radiological progression
  Using PROFILER panel (archival formalin fixed paraffin embedded tumor sample)
Optional outcome: Transcriptome | Inclusion, Day 1 cycle 2 (each cycle is 28 days), First documented radiological progression
  Using RNAseq if possible or HTG (archival formalin fixed paraffin embedded tumor sample)
Optional outcome: PBMC (in selected sites only) | Inclusion, Day 1 of cycles 2, 3, 4 and 5 (each cycle is 28 days), End of treatment plus 30 days
  Evaluation of PBMC (blood samples)
Optional outcome: ctDNA for a panel of selected genes | Inclusion, Day 1 of cycles 2, 3, 4 and 5 (each cycle is 28 days), End of treatment plus 30 days
  Evaluation of ctDNA (panel of genes to be selected at the time of analysis) (blood samples)

CONTACTS AND LOCATIONS:
Overall Officials: Jérôme FAYETTE, MD, Principal Investigator — Centre Leon Berard
Locations (17):
- France (17):
  - CHU d'Amiens, Amiens
  - ICO - Centre Paul Papin, Angers
  - Institut Sainte-Catherine, Avignon
  - Centre Georges-François Leclerc, Dijon
  - Clinique des Ormeaux, Le Havre
  - Groupe hospitalier Bretagne Sud, Lorient
  - Hôpital de la Croix-Rousse, Lyon
  - Centre Léon Bérard, Lyon
  - Hôpital de la Timone, Marseille
  - ICM - Centre Val d'Aurelle, Montpellier
  - Hôpital Privé du Confluent, Nantes
  - Centre Henri Becquerel, Rouen
  - ICO - Centre René Gauducheau, Saint-Herblain
  - Clinique Mutualiste de l'Estuaire, Saint-Nazaire
  - Centre Paul Strauss, Strasbourg
  - Institut de Cancérologie de Lorraine Alexis Vautrin, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif